CLINICAL TRIAL: NCT03714087
Title: OGS Scores After the Use of a New Finishing Protocol
Brief Title: Occlusal Outcomes by OGS After a Finishing Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Alvaro Carvajal, Professor, Universidad de Antioquia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Finishing2
Record Dates: First submitted 2018-06-04; First posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2017-06

CONDITIONS: Malocclusion; Orthodontics
Keywords: Finishing protocol; Aligner
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Intervention Model Description: One historic control group (UDEA1)comparing with intervention group (UDEA2) ( before and after)
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T1 Conventional treatment before aligner (Experimental): T1 before aligner: Conventional orthodontic treatment patients before the essix aligner
  Interventions: Device: T1 before aligner
- T2 After essix aligner (Experimental): T2 after the aligner: Essix aligner appliance with setup for 3 weeks full time
  Interventions: Other: T2 after the aligner
- Historic control group (Active Comparator): Conventional orthodontic treatment without finishing protocol UdeA2
  Interventions: Other: Historic control group

INTERVENTIONS:
Device: T1 before aligner — The UDEA2 finishing protocol include: Training of the clinicians, evaluation of finishing records, checklist according OGS items, using of aligner with set-up)
  Arms: T1 Conventional treatment before aligner
Other: T2 after the aligner — The UDEA2 finishing protocol include: Training of the clinicians, evaluation of finishing records, checklist according OGS items, using of aligner with set-up)
  Arms: T2 After essix aligner
Other: Historic control group
  Arms: Historic control group

SUMMARY:
Evaluation of the effects of the implementation of a new finishing protocol in orthodontics patients

DETAILED DESCRIPTION:
Patients who are being treated in the postgraduate orthodontic clinics and who meet the inclusion and exclusion criteria, will be subject to a detailed evaluation according to the OGS criteria and upon meeting the treatment completion criteria they will be placed an aligner with setup for 3 weeks. The scores obtained before and after the aligner will be compared with a historical control group The OGS score obtained for each group, will be compared and the impact of the protocol and the aligner will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed the active phase of the bimaxillary orthodontic treatment in the Orthodontics Postgraduate Program of the UdeA by criteria of the treating clinician, during 2014 - 2018 period were included. Patients treated by using the UDEA1 finishing protocol (GC) and the UDEA 2 (GE) finishing protocol, which included aligners. All patients must have standardized diagnostic records at the end of the finishing phase (cast models and panoramic X-Rays) and must accepted to participate in the study voluntarily

Exclusion Criteria:

* Patients that require prosthetic, periodontal and / or surgical treatments or with systemic compromise that may influence the outcome of orthodontic treatment

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
OGS score | Through study completion, an average of 2 year
  Calculation of the score of the Objective Grading System

IPD SHARING:
Plan to Share IPD: No